CLINICAL TRIAL: NCT04310267
Title: Dentoskeletal Changes Concomitant With Different Three Levels of Force Application for Maxillary Protraction in Growing Orthodontic Patients With Class 3 Malocclusion
Brief Title: Three Levels of Force Application for Maxillary Protraction
Acronym: MaxiProtr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, khaled Mohammad Taha, lecturer of orthodontics, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 345KH
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Skeletal Class 3 Malocclusion Due to Maxillary Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- classic occlusal level, low point of force application (Active Comparator): the point of force application for maxillary protraction is at the level of the occlusal plane.
  Interventions: Device: Petit typeface mask
- Nasal level, Medium point of force application (Active Comparator): the point of force application for maxillary protraction is at 20 mm from the occlusal plane (Nasal floor).
  Interventions: Device: Petit typeface mask
- Infrorbital level, High level (Active Comparator): the point of force application for maxillary protraction is at the level of the infraorbital foramen
  Interventions: Device: Petit typeface mask

INTERVENTIONS:
Device: Petit typeface mask — (Intraoral) Hyrax expander for maxilary sutures disarticulation through expansion, (Extraoral) Face mask for generating maxillary protraction forces and head gear face-bow to act as a connector between both intra and extra oral parts.
  Other Names: Hyrax expander, Head gear face-bow (Denturum)

SUMMARY:
The aim of this study is to evaluate dentoskeletal changes concomitant with different three levels of force application for maxillary protraction in growing patients with skeletal class 3 malocclusion.

DETAILED DESCRIPTION:
Nanda reported that numerous experimental studies on primates have shown orthopedic changes in response to extraoral forces; however, very few studies have made an attempt to analyze the different force variables and their relationship to facial sutures. In consideration of the variables, experimental and clinical studies were initiated in their laboratory in 1972. A study on protraction of midfacial bones on primates reported that the point of force application significantly influences the center of rotation of the maxilla in rhesus monkeys. Our unpublished data also show that centers of rotation are influenced by the magnitude of force. The study showed that the maxilla can be successfully protracted by means of carefully controlled forces.

Based on the aforementioned data, we can hypothesize that the point of force application for maxillary protraction in relation to the center of resistance of maxilla could be utilized in order to correct skeletal class 3 malocclusions with different vertical dimension discrepancies.

ELIGIBILITY:
Inclusion criteria:

The patients will be included in the study if they have the following:

1. An age range from 7 to 10 years.
2. Patients diagnosed to have skeletal class 3 malocclusion due to retruded maxilla and/or combined maxillary retrusion with mild mandibular protrusion. (based on cephalometric analysis)
3. No serious systemic diseases and/or medical treatment that could interfere with orthodontic tooth movement such as analgesics, non-steroidal anti-inflammatory drugs, and hormone supplements or antibiotics.
4. Good oral hygiene and periodontal conditions.
5. No evidence of craniofacial anomalies, such as cleft lip and palate or previous history of trauma, bruxism or parafunctions.
6. No previous orthodontic or orthognathic treatment.

Exclusion criteria:

The patients will be excluded from the study if they have the following:

1. Systemic diseases or medications that could interfere with orthodontic treatment.
2. Poor oral hygiene or periodontally compromised patients.
3. Craniofacial anomalies or previous history of trauma, bruxism or parafunctions.
4. Previous orthodontic treatment.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Amount of maxillary advancement | 8 months
  the increase in maxillary length (condalyon-A point) in mm using Cone Beam Computed Tomgraphy (CBCT)

SECONDARY OUTCOMES:
degree of maxillary rotation | 8 months
  the change in maxillary inclination (occlusal plane to SN line) in degrees using Cone Beam Computed Tomgraphy (CBCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided